CLINICAL TRIAL: NCT04569253
Title: Clinical Study to Assess the Safety and Efficacy of the Tempsure® Firm for Non-invasive Lipolysis of the Flanks.
Brief Title: Multi-Center Pivotal Study of Radiofrequency Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN20-FIRM-LIPO
Record Dates: First submitted 2020-08-27; First posted 2020-09-29 (Actual); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Body Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All study participants (Experimental): Subjects will receive treatments with the RF device on one flank. The other flank will be left untreated to serve a control.
  Interventions: Device: TempSure

INTERVENTIONS:
Device: TempSure — Non-invasive radiofrequency treatments

SUMMARY:
This is a prospective, controlled, multi-center study. Patients will be enrolled and treated with a radiofrequency device in this study if they have unwanted fat in the flank (love handle) area.

DETAILED DESCRIPTION:
Subjects are to be enrolled in this clinical study if they are 18 - 55 years old. A maximum of 55 subjects will be enrolled at up to 6 study centers. Subjects will receive up to 5 treatments with the TempSure® Firm on one flank. The other flank will be left untreated to serve a control. Subject will be required to return for follow-up visits at 6 weeks and at 12 weeks after the subject's final treatment. All subjects will receive a phone call 1 week (1-10 days) post each treatment.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female between the age of 18 - 55 years old.
* Willing to undergo treatments for fat reduction of the flank area (love handle)
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document

Exclusion Criteria:

* Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* The subject has a cut, wound, or infected skin on the area to be treated.
* The subject is on local, oral, or systemic anesthetic agents.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.
* The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months (or at the discretion of the Investigator) prior to entering this study.

Cautionary Criteria:

* The subject has any embedded electronic device that gives or receives a signal, the device should be turned off or removed prior to treatment.
* The subject has an embedded pacemaker or implantable cardioverter defibrillator (ICD), the client's cardiologist must be consulted prior to treatment.

NOTE: This device has not been tested on patients implanted with electronic devices that receive or emit signals, such as: Pacemakers, Implantable Cardiac Defibrillators (ICD), or Cardiac Resynchronization Therapy (CRT) devices.

* If the neutral pad would need to be placed on a subject that has a metal plate, rod, or any metal implant that could conduct heat from the Smart Handpiece or surgical handpiece.
* The subject is allergic to adhesives, such as glues on medical tape, they should be alerted that a rash may occur on the neutral pad site and an over the counter solution may be used to treat the area.
* The subject is allergic to gold, such as the metallic covering of the TempSure handpieces.
* The subject is allergic to corn, such as the corn derivative ingredient in Parker Aquasonic Gel.
* If the subject has an unhealthy expectation of the results - this is not plastic surgery and all subject should be fully informed of the treatment's expected results.
* The subject has nerve insensitivity to heat in the treatment area.
* The subject has severe laxity or sagging that causes redundant folds of tissue or hanging skin in the area to be treated - this treatment will be ineffective.
* The subject has used Accutane (Isotretinoin) six to twelve months prior to treatment, as this can thin the skin and make it brittle.
* Studies of the use of the RF generator on subjects that have any of the following conditions is unknown:

Autoimmune Disease Diabetic Herpes Simplex

* Use caution when treating areas that have scars, tattoos, permanent makeup, and permanent brows.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Cynosure, Inc.
Locations (6):
- United States (6):
  - Maryland Dermatology Laser, Skin, & Vein Institute, LLC., Hunt Valley, Maryland
  - JUVA Skin & Laser Center, New York, New York
  - Jeremy A Brauer MD PC, Rye, New York
  - Saluja Cosmetic and Laser Center, Huntersville, North Carolina
  - Dermatology Associates of Plymouth Meeting, P.C., Plymouth Meeting, Pennsylvania
  - McDaniel Institute of Anti-Aging Research, Virginia Beach, Virginia

REFERENCES:
- [Background] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: flanks
Period: Overall Study
Arm/Group | All Study Participants
Started | 65; 130 flanks
Control Flanks | 65; 65 flanks
Treatment Flanks | 65; 65 flanks
Completed | 57; 114 flanks
Not Completed | 8; 16 flanks

BASELINE CHARACTERISTICS:
Groups:
- RF Device Arm: Single arm, self controlled.
  TempSure: Non-invasive radiofrequency treatments
Arm/Group | RF Device Arm
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 65
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 7
  African American | 2
  Caucasian | 54
  Asian | 1
  Pacific Islander | 1
FitzPatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes used is cited in the reference section
  Participants
    Fitzpatrick Skin Type I | 1
    Fitzpatrick Skin Type II | 18
    Fitzpatrick Skin Type III | 34
    Fitzpatrick Skin Type IV | 9
    Fitzpatrick Skin Type V | 1
    Fitzpatrick Skin Type VI | 2

OUTCOME MEASURES:

1. Primary Outcome: % of Photos Identified Correctly When Comparing 12 Week Follow Up to Baseline
Description: Correct identification of pre-treatment images vs. the 12-week follow up images by blinded evaluators.
Time Frame: 12 Week Follow Up
Population: 1 subject attended the 12 week follow up so was considered complete, but did not have pictures taken for this outcome measure.
Measure: Number; unit: % of photos identified correctly
Units Other Than Participants: photographs
Groups:
- All Subject Participants: Subjects will receive treatments with the RF device on one flank. The other flank will be left untreated to serve a control.
Arm/Group | All Subject Participants
Number analyzed (Participants) | 56
Number analyzed (photographs) | 112
% of photos identified correctly | 57

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout subject participation in the study, approximately 6 months.
Description: Only subjects who received treatment on the treatment area observed adverse events (not on the control flank). Since no treatment was conducted on the control flanks, no adverse events can or should be expected for them.
Groups:
- RF Device: Subjects received treatment on this flank with the RF device.
- Control: Subjects received treatments on one flank, and their other flank (which was untreated) was used as the control. No intervention or treatment occurred on this flank.
Arm/Group | RF Device | Control
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 10/65 | 0/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RF Device (N=65) | Control (N=65)
erythema (Skin and subcutaneous tissue disorders) | 10 | 0
edema (Skin and subcutaneous tissue disorders) | 1 | 0
pain (Skin and subcutaneous tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT04569253/Prot_SAP_000.pdf